CLINICAL TRIAL: NCT01017432
Title: Compliance Of Medication After Discharge From the Hospital in the Elderly
Acronym: COMADE
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Jobin Varughese, M.D., William Beaumont Hospital
Other Study IDs: HIC 2008-252
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Compliance of Medications; Factors That May Affect Compliance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Many elderly patients have multiple medications and variable dosing regimens and the ability for hospitals to properly reconcile medications between what is given on paper to the patient and what the patients take at home depends on the patient's ability to get the medications. Some patients may delay in getting their medications from the pharmacy after being discharged. For some it may be a lack of transportation, others may feel too ill to travel and may not have family members who will be able to pick up the medications.

It is for these reasons the authors of this study want to inventory the medications that an elderly patient is being discharged on during a home visit and check on the actual prescriptions that a patient has at their house the following 1-2 days after discharge.

DETAILED DESCRIPTION:
The goal is to evaluate the effectiveness of discharge instruction in the elderly by assessing medication compliance post-discharge. Patients are identified on the units and from a Beaumont Troy discharge planning master list. Prior to discharge the patients are consented and informed they will be contacted to schedule a home visit. During the home visit, the medications the patient is currently taking are recorded. Discharge medications are recorded from the medical record following the home visit. The Investigator performing the visit is blinded to the discharge medications as the intent of the visit is only to collect data and not to ensure compliance or make clinical judgment regarding the appropriateness of the medication regimen. Anyone 65 or older can be included, who are discharged with medications and can consent. Those excluded are patients who do not live in close proximity and those discharged to extended or long-term care facilities.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients (age 65 or older)
2. Able to make own decisions (Patient has autonomy) and therefore able to make informed decisions
3. Patients with medications upon discharge from the hospital

Exclusion Criteria:

1. Patients that have the inability to give informed consent secondary to: cognitive disabilities, inability to speak or write or refusal to participate in study.
2. Patients that are younger than the age of 65.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All patients over the age of 65 who are discharged home from the hospital who meet the eligibilty criteria.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To observe compliance of medications from a discharge medication list to the meds at home after discharge from the hospital. | 18 months

SECONDARY OUTCOMES:
To observe if there are secondary factors that affect compliance (i.e. age of the patients, number of medications or herbal medications) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jobin M Varughese, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan